CLINICAL TRIAL: NCT01387958
Title: Double-blind, Randomized, Placebo-controlled, Multi-center Trial, to Determine the Safety and Antiviral Effect of 14 Days of LCQ908 Monotherapy in Hepatitis C Infected Patients
Brief Title: A Two Week Dosing Study to Determine the Safety and Antiviral Activity of LCQ908 in Hepatitis C Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to futility
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCQ908A2214
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus; Chronically infected; treatment naive; non responders to prior therapy
MeSH Terms: conditions — Hepatitis C | interventions — pradigastat

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LCQ908 (Experimental)
  Interventions: Drug: LCQ908
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCQ908
  Arms: LCQ908
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a proof of concept study, designed to look at the safety and antiviral activity of LCQ908 in hepatitis C infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male and female subjects 18 to 65 years of age with hepatitis C infections (genotypes 1, 2 or 3).
* No prior therapy or inadequate response to therapy for hepatitis C.
* Weight at least 50 kg and body mass index (BMI) within 18 - 35 kg/m2.

Exclusion Criteria:

* Use of other investigational drugs within at least 30 days of enrollment
* Women of child-bearing potential.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Measure: Change in hepatitis C viral load as assessed by PCR | 2 weeks

SECONDARY OUTCOMES:
Measure: Safety assessments will include vital signs, electrocardiograms (ECG), liver function tests, and adverse events. | 28 days
Measure: LCQ908 concentrations in the blood | over 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- New Zealand (2):
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch

REFERENCES:
- [Derived] Gane E, Stedman C, Dole K, Chen J, Meyers CD, Wiedmann B, Zhang J, Raman P, Colvin RA. A Diacylglycerol Transferase 1 Inhibitor Is a Potent Hepatitis C Antiviral in Vitro but Not in Patients in a Randomized Clinical Trial. ACS Infect Dis. 2017 Feb 10;3(2):144-151. doi: 10.1021/acsinfecdis.6b00138. Epub 2016 Nov 8. PMID 27788579